CLINICAL TRIAL: NCT03169972
Title: ADYNOVATE Drug Use-Results Survey
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 261601
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855; Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Previously treated patients (PTPs): PTPs: patients who had 4 or more days to other Factor VIII (FVIII) products
  Interventions: Biological: ADYNOVATE
- Previously untreated patients (PUPs): PUPs: patients who had 3 or less previous exposure days to other products
  Interventions: Biological: ADYNOVATE

INTERVENTIONS:
Biological: ADYNOVATE — Antihemophilic Factor (Recombinant), PEGylated
  Other Names: BAX 855; BAX855; Recombinant Factor VIII (FVIII) PEGylated

SUMMARY:
The purpose of this survey is to understand the following items in the actual clinical use of ADYNOVATE in patients:

1. Unexpected adverse drug reactions
2. Occurrence of adverse drug reactions in the actual clinical use
3. Factors that may affect safety and efficacy
4. Occurrence of Factor VIII inhibitor development in patients with coagulation factor VIII deficiency (hereinafter hemophilia A)
5. Safety and efficacy for hemophilia A patients who received routine prophylactic therapy and on-demand therapy

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A patients who receive ADYNOVATE, including previously treated patients with Factor VIII deficiency (PTPs), and previously untreated patients with Factor VIII deficiency (PUPs) who are treated with ADYNOVATE.

Exclusion Criteria:

* Patients not administered ADYNOVATE.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A (congenital blood coagulation factor VIII deficiency) who receive ADYNOVATE
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (49):
- Japan (49):
  - Nagoya City, Japan, Nagoya, Aichi-ken
  - Hirosaki City, Hirosaki, Aomori
  - Chiba-City, Japan, Chiba, Chiba
  - Matsudo City, Japan, Matsudo, Chiba
  - Narita City, Narita, Chiba
  - Matsuyama City, Japan, Matsuyama, Ehime
  - Toon City, Tōon, Ehime
  - Fukuoka-City, Japan, Fukuoka, Fukuoka
  - Kitakyusyu City, Japan, Kitakyushu, Fukuoka
  - Koriyama City, Kōriyama, Fukushima
  - Sukagawa City, Sukagawa, Fukushima
  - Ogaki City, Japan, Ōgaki, Gifu
  - Maebashi City, Maebashi, Gunma
  - Hiroshima City, Japan, Hiroshima, Hiroshima
  - Kudou-Gun, Japan, Kudou-Gun, Hokkaido
  - Sapporo City, Sapporo, Hokkaido
  - Kobe City, Kobe, Hyōgo
  - Nishinomiya City, Japan, Nishinomiya, Hyōgo
  - Morioka City, Japan, Morioka, Iwate
  - Zentuji City, Japan, Zentuji City, Kagawa-ken
  - Kagoshima City, Japan, Kagoshima, Kagoshima-ken
  - Kawasaki City, Japan, Kawasaki, Kanagawa
  - Yokohama City, Japan, Yokohama, Kanagawa
  - Koti City, Japan, Kochi, Koti Prefecture
  - Minamata City, Japan, Minamata, Kumamoto
  - Kyoto City, Kyoto, Kyoto
  - Tsu City, Japan, Tsu, Mie-ken
  - Sendai City, Sendai, Miyagi
  - Tome City, Japan, Tome, Miyagi
  - Nichinan City, Nichinan, Miyazaki
  - Matsumoto City, Matsumoto, Nagano
  - Nagano City, Japan, Nagano, Nagano
  - Jyoetsu City, Jyoetsu City, Niigata
  - Kashiwazaki City, Kashiwazaki, Niigata
  - Kurasiki City, Japan, Kurashiki, Okayama-ken
  - Okayama City, Japan, Okayama, Okayama-ken
  - Higashiosaka City, Higashiosaka, Osaka
  - Hirakata City, Hirakata, Osaka
  - Nishi-ku, Nishi-ku, Osaka
  - Osaka City, Japan, Osaka, Osaka
  - Osaka-City, Japan, Osaka, Osaka
  - Koshigaya City, Japan, Koshigaya, Saitama
  - Saitama-City, Japan, Saitama, Saitama
  - Tokushima City, Japan, Tokushima, Tokushima
  - Shinjuku-Ku, Japan, Shinjuku-Ku, Tokyo
  - Suginami-ku, Japan, Suginami-ku, Tokyo
  - Setagaya-ku, Japan, Setagaya-ku, Tokyo Metropolitan
  - Sakata City, Japan, Sakata, Yamagata
  - Shunan City, Japan, Shunan City, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc74db2bf003ab45fdb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 66 investigative sites in Japan, from 1 February 2017 to 15 September 2023.
Pre-assignment Details: Participants with a historical diagnosis of hemophilia A who received Recombinant Factor VIII (FVIII) PEGylated (ADYNOVATE) were enrolled. This included previously treated patients with Factor VIII deficiency (PTPs) and previously untreated patients with Factor VIII deficiency (PUPs) who were treated with ADYNOVATE. Participants received ADYNOVATE intravenous Infusion as part of a routine medical care.
Groups:
- Previously Treated Patients (PTPs): Participants with hemophilia A who received Recombinant Factor VIII (FVIII) PEGylated (ADYNOVATE) intravenous Infusion as part of a routine medical care. Participants in this group were previously treated patients with Factor VIII deficiency (PTPs) who had 4 or more exposure days to other Factor VIII (FVIII) products.
- Previously Untreated Patients (PUPs): Participants with hemophilia A who received Recombinant Factor VIII (FVIII) PEGylated (ADYNOVATE) intravenous Infusion as part of a routine medical care. Participants in this group were previously untreated patients with Factor VIII deficiency (PUPs) who had 3 or less previous exposure days to other Factor VIII (FVIII) products.
Period: Overall Study
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Started | 123 | 12
Completed | 123 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs) | Total
Number analyzed (Participants) | 123 | 12 | 135
Age, Customized [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    < 12 years | 29 | 6 | 35
    >= 12 years, < 18 years | 4 | 1 | 5
    >= 18 years, < 65 years | 77 | 3 | 80
    65 years or more | 7 | 2 | 9
    Unknown | 6 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 123 | 11 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 123 | 12 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 123 | 12 | 135
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 123 | 12 | 135
Healthcare Category [Count of Participants; unit: Participants]
  Inpatient | 4 | 5 | 9
  Outpatient | 119 | 7 | 126
Experience of Serious Bleeding [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Experience of Serious Bleeding | 98 | 12 | 110
    Had Experience of Serious Bleeding | 19 | 0 | 19
    Unknown | 6 | 0 | 6
Experience of Surgery [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Experience of Surgery | 91 | 9 | 100
    Had Experience of Surgery | 27 | 2 | 29
    Unknown | 5 | 1 | 6
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical History | 86 | 10 | 96
    Had Medical History | 33 | 2 | 35
    Unknown | 4 | 0 | 4
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Unknown: Data could not be collected.
  Participants
    Had No Medical Complications | 90 | 8 | 98
    Had Medical Complications | 32 | 3 | 35
    Unknown | 1 | 1 | 2
Hemophilic Arthropathy [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Hemophilic Arthropathy | 61 | 8 | 69
    Had Hemophilic Arthropathy | 60 | 3 | 63
    Unknown | 2 | 1 | 3
Target Joint of Hemophilic Arthropathy [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Target Joint of Hemophilic Arthropathy | 100 | 10 | 110
    Had Target Joint of Hemophilic Arthropathy | 17 | 0 | 17
    Unknown | 6 | 2 | 8
Hepatic Impairment [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Hepatic Impairment | 114 | 12 | 126
    Had Hepatic Impairment | 8 | 0 | 8
    Unknown | 1 | 0 | 1
Renal Impairment [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Renal Impairment | 120 | 12 | 132
    Had Renal Impairment | 2 | 0 | 2
    Unknown | 1 | 0 | 1
Allergy [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Allergy | 111 | 11 | 122
    Had Allergy | 7 | 1 | 8
    Unknown | 5 | 0 | 5
Congenital Hemophilia A [Count of Participants; unit: Participants] — Number of participants with congenital hemophilia A was reported.
  Participants | 123 | 12 | 135
Age of Diagnosis of Hemophilia A [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    < 1 year old | 38 | 3 | 41
    >= 1, < 12 years old | 28 | 3 | 31
    <=18 years | 3 | 1 | 4
    >= 18, < 65 years old | 4 | 3 | 7
    >= 65 years old | 1 | 1 | 2
    Unknown | 49 | 1 | 50
Times of Bleeding in One Year [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    < 1 time per a year | 29 | 4 | 33
    >= 1, < 10 times per a year | 44 | 0 | 44
    >= 10 times per a year | 14 | 0 | 14
    Unknown | 36 | 8 | 44
Severity of Hemophilia A [Count of Participants; unit: Participants] — Number of participants in each category of severity of hemophilia A was reported. Severity of hemophilia A was categorized as Severe (Factor VIII activity was less than 1%), Moderate (1~5%), and Mild (5% or more). Unknown: Data could not be collected.
  Participants
    Severe | 93 | 8 | 101
    Moderate | 16 | 2 | 18
    Mild | 7 | 2 | 9
    Unknown | 7 | 0 | 7
Dosing Regimen before the Start of Administration of ADYNOVATE [Count of Participants; unit: Participants] — Number of participants with regimens before the start of administration of ADYNOVATE were reported (Prophylaxis Therapy, On-demand Replacement Therapy, Prophylaxis and On-demand Replacement Therapy, The Other Therapy, and Had Not Treated). Had Not Treated: Participants in this category had not been received any does for hemophilia A before the start of administration of ADYNOVATE.
  Participants
    Prophylaxis Therapy | 78 | 0 | 78
    On-demand Replacement Therapy | 21 | 4 | 25
    Prophylaxis and On-demand Replacement Therapy | 22 | 0 | 22
    The Other Therapy | 2 | 1 | 3
    Had Not Treated | 0 | 7 | 7
Factor VIII Inhibitor Development [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Factor VIII Inhibitor Development | 97 | 7 | 104
    Had Factor VIII Inhibitor Development | 7 | 0 | 7
    Unknown | 19 | 5 | 24
Family History of Hemophilia [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Family History of Hemophilia | 52 | 4 | 56
    Had Family History of Hemophilia | 46 | 5 | 51
    Unknown | 25 | 3 | 28
Family History of Inhibitor Development [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Had No Family History of Inhibitor Development | 85 | 5 | 90
    Had Family History of Inhibitor Development | 6 | 0 | 6
    Unknown | 32 | 7 | 39
Status of Concomitant Drugs [Count of Participants; unit: Participants] — Number of participants who received concomitant drugs at the start of this survey was reported.
  Participants | 34 | 7 | 41
Status of Concomitant Therapies [Count of Participants; unit: Participants] — Number of participants who received concomitant therapies at the start of this survey was reported.
  Participants | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued the Use of Study Drug
Description: Number of previously treated patients (PTPs) and previously untreated patients (PUPs) who discontinued the use of ADYNOVATE were reported.
Time Frame: Throughout the study participation period: 1 year for previously treated patients for PTPs and 2 years for previously untreated patients for PUPs
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 123 | 12
Participants | 10 | 5

2. Primary Outcome: Annual Bleed Rate (ABR) of Spontaneous Bleeding Episodes on a Prophylaxis Regimen
Description: Annual bleed rate (ABR) of spontaneous bleeding episodes in PTPs and PUPs on a prophylaxis regimen were reported. Annual bleed rate is calculated by the number of bleeding episodes observed during administration period divided by the duration of administration period, after that multiplied with 365.2425.
Time Frame: as for outcome 1
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis who treated with a prophylaxis regimen and experienced spontaneous bleeding episodes during the administration period.
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 24 | 0
Bleeds per year | 1.99 [1.00 to 3.59] |

3. Primary Outcome: Annual Bleed Rate (ABR) of Breakthrough Bleeding Episodes on a Prophylaxis Regimen
Description: Annual bleed rate (ABR) of breakthrough bleeding episodes in PTPs and PUPs on a prophylaxis regimen were reported. Annual bleed rate is calculated by the number of bleeding episodes observed during administration period divided by the duration of administration period, after that multiplied with 365.2425.
Time Frame: as for outcome 1
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis who treated with a prophylaxis regimen and experienced breakthrough bleeding episodes during the administration period.
Measure: Median (Inter-Quartile Range); unit: Bleeds per year
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 31 | 1
Bleeds per year | 3.16 [1.11 to 5.10] | 2.91 [2.91 to 2.91]

4. Primary Outcome: Duration of Treatment of Study Drug on a Prophylaxis Regimen
Description: Duration of treatment of study drug on a prophylaxis regimen was reported.
Time Frame: as for outcome 1
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed was the number of participants with data available for analysis who treated with a prophylaxis regimen during the administration period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 110 | 7
days | 343.0 (69.33) | 510.7 (256.04)

5. Primary Outcome: Duration of Treatment of Study Drug an On-Demand Regimen
Description: Duration of treatment of study drug on an on-demand regimen was reported.
Time Frame: as for outcome 1
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed was the number of participants with data available for analysis who treated with an on-demand regimen during the administration period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 14 | 3
days | 13.3 (22.42) | 5.0 (2.65)

6. Primary Outcome: Dose Per Administration of Study Drug on a Prophylaxis Regimen
Description: Dose per administration of study drug on a prophylaxis regimen was reported.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU per kilograms (kg)
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 110 | 7
IU per kilograms (kg) | 39.4 (12.69) | 45.8 (7.70)

7. Primary Outcome: Dose Per Administration of Study Drug an On-Demand Regimen
Description: Dose per administration of study drug on an on-demand regimen was reported.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: IU per kilograms (kg)
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 14 | 3
IU per kilograms (kg) | 36.8 (13.88) | 29.7 (12.42)

8. Secondary Outcome: Number of Doses Per a Week of Study Drug on a Prophylaxis Regimen
Description: Number of doses per a week of study drug on a prophylaxis regimen was reported.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Number of doses per a week
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 110 | 7
Number of doses per a week | 2.0 (0.38) | 1.8 (0.41)

9. Primary Outcome: Number of Doses Per a Bleeding Episode of Study Drug an On-Demand Regimen
Description: Number of doses per a bleeding episode of study drug on an on-demand regimen was reported.
Time Frame: as for outcome 1
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis who treated with an on-demand regimen during the administration period.
Measure: Mean (Standard Deviation); unit: Number of doses per a bleeding episode
Units Other Than Participants: Count of Bleeding Episodes
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 14 | 3
Number analyzed (Count of Bleeding Episodes) | 58 | 3
Number of doses per a bleeding episode | 6.0 (4.45) | 5.0 (4.36)

10. Primary Outcome: Hemostatic Effectiveness of Study Drug on Treatment of Breakthrough Bleeding Episodes With a Prophylaxis Regimen
Description: Percentage of each category of hemostatic effectiveness for treatment of breakthrough bleeding episodes in a prophylaxis regimen assessed by the investigator was reported. Hemostatic effectiveness was assessed by the investigator with following 4-point ordinal scale: Excellent, Good, Fair, Poor.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Percentage of bleeding episodes
Units Other Than Participants: Count of Bleeding Episodes
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 32 | 3
Number analyzed (Count of Bleeding Episodes) | 86 | 5
Percentage of bleeding episodes
  Excellent | 37.21 | 20.00
  Good | 62.79 | 40.00
  Fair | 0.00 | 0.00
  Poor | 0.00 | 20.00

11. Primary Outcome: Hemostatic Effectiveness of Study Drug on an On-Demand Regimen
Description: Percentage of each category of hemostatic effectiveness for an on-demand regimen assessed by the investigator was reported. Hemostatic effectiveness was assessed by the investigator with following 4-point ordinal scale: Excellent, Good, Fair, Poor.
Time Frame: as for outcome 1
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey. The number analyzed was the number of participants with data available for analysis who treated with on-demand regimen during the administration period.
Measure: Number; unit: Percentage of bleeding episodes
Units Other Than Participants: Count of Bleeding Episodes
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 14 | 3
Number analyzed (Count of Bleeding Episodes) | 58 | 3
Percentage of bleeding episodes
  Excellent | 32.76 | 33.33
  Good | 60.34 | 33.33
  Fair | 6.90 | 0.00
  Poor | 0.00 | 33.33

12. Secondary Outcome: Number of Participants Who Experience Factor VIII Inhibition, Dermatitis Atopic or Eczema as an Adverse Event (AE)
Description: Number of PTPs and PUPs who experienced factor VIII inhibition, dermatitis atopic or eczema as an AE related to development of inhibitors, shock or anaphylaxis was reported.
Time Frame: as for outcome 1
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
Number analyzed (Participants) | 123 | 12
Participants
  Factor VIII Inhibition | 1 | 3
  Dermatitis Atopic | 0 | 1
  Eczema | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 1 year for previously treated patients (PTPs) or up to 2 years for previously untreated patients (PUPs)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Previously Treated Patients (PTPs) | Previously Untreated Patients (PUPs)
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/123 | 1/12
Other Adverse Events (participants affected / at risk) | 1/123 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Previously Treated Patients (PTPs) (N=123) | Previously Untreated Patients (PUPs) (N=12)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Factor VIII inhibition (Blood and lymphatic system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previously Treated Patients (PTPs) (N=123) | Previously Untreated Patients (PUPs) (N=12)
Nasopharyngitis (Infections and infestations) | 0 | 1
Factor VIII inhibition (Blood and lymphatic system disorders) | 1 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT03169972/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT03169972/SAP_001.pdf